CLINICAL TRIAL: NCT04511403
Title: Prevalence of Oral Mucosal Alterations In a Sample of Egyptian Patients With Cardiovascular Diseases: A Hospital- Based Cross-Sectional Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abd El Basset Mostafa Mohamed Sleem, Principle investigator, Cairo University
Other Study IDs: Mucosal changes
Record Dates: First submitted 2020-08-08; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
to assess the oral mucosal alterations and their prevalence secondary to use cardiovascular drugs in a sample of Egyptian population with cardiovascular diseases .

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) still a major cause of health loss for all regions of the world. Sociodemographic change over the past 25 years has been associated with the dramatic decrease in CVD in regions with very high sociodemographic index (SDI), but only a gradual decrease or no change in most regions (Roth et al., 2017).

Statistics from the World Health Organization indicates that cardiovascular diseases are the leading cause of death in Egypt, accounting for 46% of total deaths ( Royal Philips,2018).

The mouth serves as "a mirror of health or disease, as a sentinel or early warning system, as an accessible model for the study of other tissues and organs, and as a potential source of pathology affecting other systems and organs (Dr. Shantala Arunkumar, 2013).

The oral cavity is considered as a window to the body because oral manifestations accompany many systemic diseases. In many instances, oral involvement first appears than other symptoms or lesions at other locations. These oral manifestations must be properly recognized if the patient is to receive appropriate diagnosis and referral for treatment (Mehrotra et al., 2010b).

People with cardiovascular disease and who are at high cardiovascular risk (due to the presence of one or more risk factors such as hypertension, diabetes, hyperlipidaemia or already established disease) need early detection and management using counselling and medicines, as appropriate(World Health Organization, 2013).

A great many cardiovascular drugs have adverse reactions in the mouth in the form of xerostomia, lichenoid reactions, burning mouth sensation, loss of taste sensation, gingival hyperplasia and bleeding(Arunkumar, 2013).

Cardiovascular disease is the main cause of early death among people with diabetes. People with diabetes also suffer from hypertension, dyslipidaemia, and obesity, which contribute to increased incidence of cardiovascular disease (Malik and Dwivedi, 2015).

CVDs are a leading cause of death worldwide including the Middle East. This is caused in part by the dysregulation of adipose tissue cause increasing in production of pro-inflammatory adipokines and reduction in cardio-protective adipokines such as adiponectin (Abu-Farha, Behbehani and Elkum, 2014).

Low- and middle-income countries are disproportionally affected: over 80% of CVD deaths take place in low- and middle-income countries and occur almost equally in men and women. By 2030, almost 23.6 million people will die from CVDs, mainly from heart disease and stroke (WHO, 2015).

Medications used for management of hypertension cause oral alternation like Diuretics cause oral dryness, adrenergic inhibitors cause oral dryness and ulcerations, calcium antagonists cause overgrowth of gingiva while ACE inhibitors affect test sensation and lichenoid reactions of the oral mucosa (Mehrotra et al., 2010).

ELIGIBILITY:
Inclusion Criteria:

* 1-Patients >18-years-old. 2-Patients diagnosed with cardiovascular diseases (Ivanuša, 2014). 3-patients taking cardiovascular drugs(Dr. Shantala Arunkumar, 2013).

Exclusion Criteria:

* 1- Patients not physically able to participate in survey or clinical oral examination.

  2- Patients under immunosuppressive drugs. 3-Patients with dementia or confusion, severe illness. 4- patients who refuse to participate in the study. 5-patients with hormonal diseases like diabetes mellitus and others. 6-patients with conditions cause xerostomia like Sjogren's syndrome and any medical diseases other than cardiovascular diseases.

  7-patients suffering from any medical diseases with aphthous ulcer and any other cause of xerostomia than cardiovascular diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital- Based Cross-Sectional Study
Sampling Method: Non-Probability Sample
Enrollment: 338 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Oral mucosal manifestations as listed (Dr. Shantala Arunkumar, 2013) | through study completion, an average of 1 year
  Clinical examination according to WHO (World Health Organization, 2010) Oral mucosal manifestations as listed (Dr. Shantala Arunkumar, 2013) Clinical examination according to WHO (World Health Organization, 2010) Dichotomous outcome (Yes/No).

SECONDARY OUTCOMES:
Periodontal condition.(Miranda et al., 2012) | through study completion, an average of 1 year
  Clinical examination with GO-index(Normal- Mild ≤2 -Moderate 2-4 mm- sever≥4 mm)
Salivary glands function | through study completion, an average of 1 year
  Clinical oral dryness examination (Jager et al., 2018) in addition using Xerostomia questionnaire (Wiener et al., 2010)

REFERENCES:
- [Background] Abu-Farha M, Behbehani K, Elkum N. Comprehensive analysis of circulating adipokines and hsCRP association with cardiovascular disease risk factors and metabolic syndrome in Arabs. Cardiovasc Diabetol. 2014 Apr 9;13:76. doi: 10.1186/1475-2840-13-76. PMID 24716628
- [Background] Jager DHJ, Bots CP, Forouzanfar T, Brand HS. Clinical oral dryness score: evaluation of a new screening method for oral dryness. Odontology. 2018 Oct;106(4):439-444. doi: 10.1007/s10266-018-0339-4. Epub 2018 Jan 22. PMID 29356914
- [Background] Habbab KM, Moles DR, Porter SR. Potential oral manifestations of cardiovascular drugs. Oral Dis. 2010 Nov;16(8):769-73. doi: 10.1111/j.1601-0825.2010.01686.x. PMID 20604876